CLINICAL TRIAL: NCT00004932
Title: A Phase I Study of STI571 in Ph+ Leukemia
Brief Title: STI571 in Treating Patients With Recurrent Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P9973; COG-P9973 (Other: Children's Oncology Group); POG-9973 (Other: Pediatric Oncology Group); CCG-P9973 (Other: Children's Cancer Group); CDR0000067616 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 260 mg/m2 imatinib mesylate (ST571) (Experimental)
  Interventions: Drug: imatinib mesylate
- 340 mg/m2 imatinib mesylate (ST571) (Experimental)
  Interventions: Drug: imatinib mesylate
- 440 mg/m2 imatinib mesylate (ST571) (Experimental)
  Interventions: Drug: imatinib mesylate
- 570 mg/m2 imatinib mesylate (ST571) (Experimental)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate
  Other Names: CGP 57148; IND # 55666

SUMMARY:
RATIONALE: Imatinib mesylate may interfere with the growth of cancer cells and may be an effective treatment for leukemia.

PURPOSE: Phase I trial to study the effectiveness of imatinib mesylate in treating patients who have recurrent leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of imatinib mesylate in patients with recurrent Philadelphia chromosome-positive leukemia.
* Characterize the pharmacokinetic behavior of this drug in this patient population.
* Determine preliminarily the antileukemic activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral imatinib mesylate (STI571) once daily for 28 days. Treatment continues in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of STI571 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 32 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Recurrent Philadelphia (Ph) chromosome-positive leukemia

  * Recurrent or refractory acute lymphoblastic or myeloblastic leukemia OR
  * Chronic myelogenous leukemia with resistance to interferon alfa with any of the following:

    * WBC at least 20,000/mm^3 after at least 3 months of interferon therapy
    * At least 100% increase in WBC to at least 20,000/mm^3 confirmed over 2 weeks while receiving interferon alfa
    * At least 66% Ph chromosome-positive cells after 1 year of interferon therapy
    * At least 30% increase in number of Ph chromosome-positive cells after an interferon-induced response while continuing interferon therapy

PATIENT CHARACTERISTICS:

Age:

* Under 22

Performance status:

* Karnofsky 50-100% if over 10 years of age OR
* Lansky 50-100% if 10 years of age and under

Life expectancy:

* At least 8 weeks

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGPT less than 3 times normal
* Albumin greater than 2 g/dL

Renal:

* Creatinine no greater than 1.5 times normal OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* If prior allogeneic stem cell transplantation, no uncontrolled graft-versus -host disease
* No seizure disorder if on anticonvulsants
* No uncontrolled infection
* No CNS toxicity greater than grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 1 week since prior biologic therapy and recovered
* At least 3 months since prior stem cell transplantation (SCT)
* At least 1 week since prior growth factors
* At least 1 week since prior interferon alfa

Chemotherapy:

* Recovered from prior chemotherapy
* At least 6 weeks since prior busulfan and nitrosoureas
* At least 2 weeks since prior homoharringtonine
* At least 1 week since low-dose cytarabine
* At least 2 weeks since prior moderate-dose cytarabine
* At least 4 weeks since prior high-dose cytarabine
* At least 3 weeks since all other prior cytotoxic chemotherapies
* No prior hydroxyurea

Endocrine therapy:

* Must be on a stable dose of steroids if received prior allogeneic SCT

Radiotherapy:

* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior craniospinal radiotherapy
* At least 6 months since prior radiotherapy to 50% or more of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational agents
* No concurrent anticonvulsants

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2002-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Survival | Length of study
  To estimate the maximum tolerated dose (MTD) of STI571 administered orally once daily without interruption to children with recurrent Ph+ leukemia.

SECONDARY OUTCOMES:
Dose-limiting toxicities | Length of study
  To determine the dose-limiting toxicities (DLT) of STI571 given on this schedule.
Characterize the pharmacokinetic behavior | Length of study
  To characterize the pharmacokinetic behavior of STI571 in children with recurrent Ph+ leukemia.
Define the anti-leukemic activity of STI571 | Length of study
  To preliminarily define the anti-leukemic activity of STI571 within the confines of a Phase I study.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Champagne, MD, Study Chair — Hopital Sainte Justine
Locations (235):
- United States (206):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Childhood Hematology/Oncology Associates, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. Dupont Institute, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami-Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Inc., Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Raymond Blank Memorial Hospital for Children, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's/Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Atlantic Health System, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - State University of New York Health Science Center at Brooklyn College of Medicine, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Doernbecher Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at JCMC, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Health Care System, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Charleston, Charleston, West Virginia
  - Cabell-Huntington Hospital, Inc, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Laval University Medical Center, Sainte-Foy, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Result] Champagne MA, Capdeville R, Krailo M, Qu W, Peng B, Rosamilia M, Therrien M, Zoellner U, Blaney SM, Bernstein M; Children's Oncology Group phase 1 study. Imatinib mesylate (STI571) for treatment of children with Philadelphia chromosome-positive leukemia: results from a Children's Oncology Group phase 1 study. Blood. 2004 Nov 1;104(9):2655-60. doi: 10.1182/blood-2003-09-3032. Epub 2004 Jul 1. PMID 15231574
- [Result] Champagne MA, Hershon L, Rosamilia M, et al.: STI571 in the Treatment of Pediatric Philadelphia (Ph+) Chromosome-Positive Leukemia: A Children's Oncology Group Phase 1 Study (P-9973). [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1466, 2001.